CLINICAL TRIAL: NCT04035681
Title: Stroke Survivor-Caregiver Dyads: Feasibility of a Brief Psychosocial Intervention for Depressive Symptoms and Quality of Life
Brief Title: Problem-Solving Therapy for Depressive Symptoms and Quality of Life in Stroke Survivor-Caregiver Dyads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Collaborators: University of Minnesota (Other); Agnes Marshall Walker Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1368980-3
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Quality of Life; Depression
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem-Solving Therapy (Experimental): Participants who are assigned to receive problem-solving therapy will work with a research team member for six, one-hour sessions. During each session, participants will identify a problem (big or small) and create a plan to work on that problem.
  Interventions: Behavioral: Problem-Solving Therapy
- Stroke-Related Health Education (Active Comparator): Participants who are assigned to receive stroke-related health education will work with a research team member who will teach them about various topics related to stroke over six, one-hour sessions. Each session will cover information about a different topic related to stroke.
  Interventions: Other: Stroke-Related Health Education

INTERVENTIONS:
Behavioral: Problem-Solving Therapy — Problem-Solving Therapy is a brief psychosocial intervention for management of depressive symptoms. Participants will have six, one-hour sessions with an interventionist to learn a structured approach to problem-solving.
  Arms: Problem-Solving Therapy
Other: Stroke-Related Health Education — The stroke-related health education program will teach participants about various topics related to stroke. Participants will have six, one-hour sessions with an interventionist to learn about different topics related to stroke.
  Arms: Stroke-Related Health Education

SUMMARY:
The purpose of this feasibility study is to determine whether it is practical and helpful to provide problem-solving therapy to stroke survivors and their spouses/partners (caregivers) together. It will also compare the experiences of participants who receive problem-solving therapy to those who receive stroke-related health education.

Many stroke survivors and caregivers report feeling sad or blue at some point after the stroke. These feelings can impact quality of life. Encountering problems is a part of daily life. These problems can be big or small, but sometimes they can pile up and feel overwhelming, contributing to feelings of sadness. Problem-solving therapy is a tool that teaches structured ways to address current problems or challenges in your life.

Participants who are assigned to receive problem-solving therapy will work with a research team member for six, one-hour sessions. During each session, participants will identify a problem (big or small) and create a plan to work on that problem.

Participants who are assigned to receive stroke-related health education will work with a research team member who will teach them about various topics related to stroke over six, one-hour sessions. Each session will cover information about a different topic related to stroke.

Outcomes data will be collected at approximately 4 weeks, 8 weeks, and 13 weeks from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Both dyad participants are at least 18 years of age.
2. The stroke survivor experienced an ischemic or hemorrhagic stroke at least 3 months prior to enrollment.
3. The caregiver is a spouse/partner who provides regular, unpaid support for the survivor in activities of daily living.
4. Both dyad members are willing and able understand and comply with protocol requirements.

Exclusion Criteria:

1. The stroke survivor has severe expressive or receptive aphasia or global aphasia, as documented in the medical record by a speech pathologist or other provider.
2. Either dyad member is unable to write, as this will interfere with completion of MiniCog assessment.
3. Either dyad member has significant cognitive impairment, evidenced by MiniCog score <4 at screening.
4. Either dyad member reports an intent to harm him/herself or others.
5. Either dyad member has any concurrent conditions that would interfere with participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Study Retention | Through study completion, an average of 13 weeks.
  Total percentage of participants who complete the study.
Protocol Adherence | Through study completion, an average of 13 weeks.
  Total percentage of protocol-specified activities completed by enrolled participants.
Intervention Acceptability | Post-intervention, at approximately 8 weeks.
  Participant experience collected via self-report survey.
Study Recruitment Success | At initial contact.
  Percentage of eligible candidates who enroll in the study.

SECONDARY OUTCOMES:
Pre/post-intervention changes in depressive symptoms among caregivers. | Baseline and post-intervention, covering an average of 8 weeks.
  Pre/post-intervention changes in 9-item Patient Health Questionnaire (PHQ-9) scores.
Pre/post-intervention changes in quality of life among caregivers. | Baseline and post-intervention, covering an average of 8 weeks.
  Pre/post-intervention changes in Euroqol 5-item QOL scale (EQ-5D) scores.
Pre/post-intervention changes in depressive symptoms among stoke survivors. | Baseline and post-intervention, covering an average of 8 weeks.
  Pre/post-intervention changes in 9-item Patient Health Questionnaire (PHQ-9) scores.
Pre/post-intervention changes in quality of life among stoke survivors. | Baseline and post-intervention, covering an average of 8 weeks.
  Pre/post-intervention changes in Euroqol 5-item QOL scale (EQ-5D) scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Allina Health, Minneapolis, Minnesota, United States